CLINICAL TRIAL: NCT05970445
Title: Clinical Phenotypic Characteristics of the Solute Carrier Family 26 Member 4 (SC26A4) Mutation in Pendred Syndrome/Nonsyndromic Enlarged Vestibular Aqueduct (PS/NSEVA)
Brief Title: Clinical Phenotypic Characteristics of SC26A4
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Shiming Yang, PhD, Departmant of Otolaryngology Head and Neck Surgery, Chinese PLA General Hospital
Other Study IDs: PS/NSEVA-01
Record Dates: First submitted 2023-06-12; First posted 2023-08-01 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Hearing Loss; Pendred Syndrome
MeSH Terms: conditions — Hearing Loss; Pendred syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — SLC26A4 sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with enlarged vestibular aqueduct: This study will analyze the SLC26A4 mutation, and audiological and imaging characteristics of PS/NSEVA to summarize the clinical manifestations of PS/NSEVA patients. The study also will analyze the effects of SLC26A4 mutation and inner ear imaging on the degree of hearing loss in PS/NSEVA patients to provide predictive measures for the genetic diagnosis and clinical phenotype of PS/NSEVA. Finally, the effects of sex and age on the degree of hearing loss in patients with PS/NSEVA will be analyzed to provide insight on PS/NSEVA pathogenesis.

SUMMARY:
The presence or absence of SC26A4, whether combined with Mondini malformation, and patient age, are important factors affecting the degree of hearing loss in the Chinese population.

DETAILED DESCRIPTION:
To summarize the Solute Carrier Family 26 Member 4 (SLC26A4) mutation and clinical phenotypic characteristics of Pendred Syndrome/Nonsyndromic Enlarged Vestibular Aqueduct (PS/NSEVA) patients and provide evidence supporting the clinical diagnosis and genetic counseling of patients with PS/NSEVA. A retrospective cohort study for the Chinese population is needed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Enlarged Vestibular Aqueduct;
2. Patients with hearing loss;
3. Patients with results of SLC26A4 sequencing;

Exclusion Criteria:

Subjects will be excluded from this study if any of the following are present:

1. Audiometric data is incomplete
2. Incomplete basic information
3. Patients who did not undergo HRCT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Because the influencing factors and pathological mechanisms of PS/NSEVA patients are intricate, there are many controversies regarding the relationship between the SLC26A4 gene, the degree of hearing loss experienced by PS/NSEVA patients, and the relationship between inner ear imaging and audiology.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
SLC26A4 sequencing | through study completion, an average of 0.5 year
  Extraction from patient clinical information database and secondary use. From each patient included in the study, 3 ml of peripheral blood was collected and the DNA extracted for the diagonosis in the past.
High-resolution computed tomography of the temporal bone | through study completion, an average of 0.5 year
  Extraction from patient clinical information database and secondary use. High-resolution computed tomography of the temporal bone is used to measure the width of the vestibular aqueduct (VA) in the left and right ears to determine whether other inner ear malformations exist.
Hearing test | through study completion, an average of 0.5 year
  Extraction from patient clinical information database and secondary use. The Auditory Steady State Response test is conducted to evaluate the degree of hearing loss.

CONTACTS AND LOCATIONS:
Overall Officials: Shiming Yang, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China